CLINICAL TRIAL: NCT07247292
Title: A Multicenter Non-interventional Single-arm Retrospective-prospective Observational Study in Therapeutic Approaches on AQP4-IgG Positive Neuromyelitis Optica Spectrum Disorder (NMOSD) in Real Clinical Practice in Russia
Brief Title: Epidemiological Study of Treatment Approaches on AQP4-IgG Positive NMOSD in Russia
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D9282R00001
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Rare Diseases; Neuromyelitis Optica Spectrum Disorder (NMOSD)
MeSH Terms: conditions — Rare Diseases; Neuromyelitis Optica

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

SUMMARY:
This is a multi-centre, retrospective-prospective, single-arm, non-interventional (observational) cohort study with secondary data collection within real-world settings of participants with AQP4-IgG positive NMOSD.

DETAILED DESCRIPTION:
This is a multicenter, retrospective-prospective, single-arm observational cohort study using secondary data collection from routine care medical records.

The primary objective is to describe baseline demographic and clinical characteristics, diagnostic algorithms, and treatment approaches. Secondary objectives are to describe Expanded Disability Status Scale (EDSS) levels and dynamics, collect the rate, duration, and reasons for hospitalizations, and evaluate physician-reported relapse profiles.

Approximately 100 adults will be enrolled consecutively across about 10 specialized sites. The study will sequentially include only those patients who have signed the informed consent form (ICF). Eligible patients will be enrolled consecutively at each site to minimize selection bias. Each participant will be followed for 36 months from informed consent (T0), with data collection every 6 months (T1-T6). The baseline period is defined as the time from NMOSD diagnosis until inclusion, with retrospective data abstraction; subsequent data are collected prospectively at routine visits. All data are entered into an electronic case report form (eCRF) from paper/electronic medical records. No study-specific interventions are performed; treatment is determined by usual care.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (≥18 years) with a confirmed diagnosis of AQP4-IgG positive NMOSD following the 2015 IPND criteria;
2. Provision of signed and dated written informed consent.

Exclusion Criteria:

1.Participants currently enrolled in clinical studies for the treatment of NMOSD.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants of both sexes aged 18 years and older with diagnosis of AQP4-IgG positive NMOSD established according to 2015 IPND criteria will be enrolled in various clinical institutions in Russia that provide treatment for NMOSD patients.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-12-23 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Baseline demographics and clinical characteristics | At inclusion
  Summary of participant demographics and clinical history at inclusion: age at inclusion and at NMOSD diagnosis, sex, ethnicity, BMI at inclusion, disease duration, clinical symptoms at inclusion, comorbidities.
Pre-inclusion relapse history | From NMOSD diagnosis to inclusion (retrospective baseline)
  Proportion of patients with ≥1 and >1 physician-reported relapses and severe relapses (EDSS increase ≥2.0 points from baseline per event); annualized relapse rate (ARR) prior to inclusion.
Pre-inclusion NMOSD-related hospitalizations | From NMOSD diagnosis to inclusion (retrospective baseline)
  Number of patients with NMOSD-related hospitalizations from the time of NMOSD diagnosis; median cumulative duration (days) of NMOSD-related hospitalizations prior to inclusion.
Time from first symptoms to NMOSD diagnosis | From first NMOSD symptoms to date of diagnosis (retrospective baseline)
  Median time (months) from patient-reported first NMOSD symptoms to confirmed NMOSD diagnosis according to 2015 IPND criteria.
Prior misdiagnoses profile | From first NMOSD symptoms to confirmed NMOSD diagnosis (retrospective baseline)
  Proportion of patients with any prior misdiagnosis and by type (e.g., MS, MOGAD, CNS infections, SLE only, Sjögren's only, Behçet's, neurosarcoidosis, CNS vascular disease, toxic/metabolic, neoplasms/paraneoplastic, congenital CNS, other).
AQP4-IgG testing method | At time of NMOSD diagnostic workup (retrospective baseline)
  Number and proportion of patients tested by cell-based assay versus ELISA for AQP4-IgG serostatus determination.
MRI brain T2-hyperintense lesion count change | Baseline (≤12 months pre-inclusion) and Months 6, 12, 18, 24, 30, and 36 post-inclusion
  Mean change from baseline in the number of T2-hyperintense brain lesions; presence of T1 contrast-enhancing lesions recorded as categorical variables.
Optic nerve MRI findings | Baseline (≤12 months pre-inclusion) and Months 6, 12, 18, 24, 30, and 36 post-inclusion
  Presence of contiguous lesions, bilateral neuritis, chiasmal extension, and optic nerve atrophy recorded as categorical variables per timepoint.
Spinal cord MRI lesion metrics | Baseline (≤12 months pre-inclusion) and Months 6, 12, 18, 24, 30, and 36 post-inclusion
  T2 lesion count; presence of longitudinally extensive lesions (≥3 segments), transverse lesions, and spinal cord atrophy extending ≥3 segments recorded as categorical variables per timepoint.
Relapse prevention therapy patterns | From NMOSD diagnosis to inclusion and Months 6, 12, 18, 24, 30, and 36 post-inclusion
  Number of patients receiving relapse prevention therapy by regimen: immunosuppressive drugs monotherapy; biologic monotherapy; biologic plus immunosuppressive combination; mean daily corticosteroid dose if low-dose steroids used (prednisolone-equivalent).
Acute relapse treatment modalities | From NMOSD diagnosis to inclusion and Months 6, 12, 18, 24, 30, and 36 post-inclusion
  Number of patients receiving high-dose corticosteroids, plasma exchange, or immunoadsorption for acute relapses; summarized per period.
Concomitant medications | From NMOSD diagnosis to inclusion and Months 6, 12, 18, 24, 30, and 36 post-inclusion
  Number of patients by class/type of concomitant medications for comorbid conditions recorded from diagnosis to inclusion and prospectively.

SECONDARY OUTCOMES:
EDSS mean at each time point | Baseline (T0) and Months 6 (T1), 12 (T2), 18 (T3), 24 (T4), 30 (T5), 36 (T6)
  Expanded Disability Status Scale (EDSS) mean score across participants at each scheduled assessment; EDSS assessed per routine clinical practice.
EDSS mean change from baseline | Months 6 (T1), 12 (T2), 18 (T3), 24 (T4), 30 (T5), 36 (T6)
  Mean change in EDSS from baseline (T0) to each follow-up time point; change calculated as EDSS at time point minus baseline EDSS.
All-cause hospitalizations | From inclusion (T0) through Month 36 (T6)
  Number of patients with ≥1 hospitalization from any cause during follow-up; counts summarized overall and by hospitalization cause categories.
Median cumulative duration of hospitalizations | From inclusion (T0) through Month 36 (T6)
  Median cumulative number of days spent hospitalized per patient during follow-up; calculated across all hospitalizations per participant.
NMOSD-related hospitalizations | From inclusion (T0) through Month 36 (T6)
  Number of patients with ≥1 hospitalization due to NMOSD during follow-up; NMOSD-related as documented in medical records.
Median cumulative duration of NMOSD-related hospitalizations | From inclusion (T0) through Month 36 (T6)
  Median cumulative number of days spent hospitalized per patient for NMOSD-related causes during follow-up.
Patients with physician-reported relapse(s) | From inclusion (T0) through Month 36 (T6)
  Number of patients with ≥1 and >1 physician-reported NMOSD relapse during follow-up; relapses defined per protocol and documented by clinician assessment.
Patients with severe relapse(s) | From inclusion (T0) through Month 36 (T6)
  Number of patients with ≥1 and >1 severe NMOSD relapse during follow-up; severe relapse defined as EDSS increase ≥2.0 points from baseline (for myelitis) or major OSIS exacerbation, per protocol.
Annualized relapse rate (ARR) | From inclusion (T0) through Month 36 (T6)
  ARR calculated as total number of physician-reported relapses divided by person-years observed during follow-up for each patient, summarized at the cohort level.
Median time to first physician-reported relapse | From inclusion (T0) to first relapse event, up to Month 36 (T6)
  Time from inclusion (T0) to first physician-reported NMOSD relapse; analyzed using Kaplan-Meier methods with censoring at Month 36 or withdrawal.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Novosibirsk, Russia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/